CLINICAL TRIAL: NCT05677204
Title: Factors Predicting the Course of Acute Achilles Tendinopathy in Runners
Brief Title: Influencing Factors of Acute Achilles Tendinopathy in Runners
Acronym: AchTend
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Principal Investigator, Laval University
Other Study IDs: 2021-2162, _RIS
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Achilles Tendinopathy
Keywords: Runners; Acute; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Achilles tendinopathy: No intervention will be given

SUMMARY:
Achilles tendinopathy is highly prevalent in runners, but its evolution is not easily predictable. The aim of this study is to evaluate the impact of clinical and social factors on the prognosis of acute (less than 3 months) Achilles tendinopathy in runners. Runners will be evaluated in person twice. At their first visit, data related to their training (frequency, intensity, …), their running pattern (cadence, foot contact angle) and shoes (minimalist index) will be collected. Moreover, an ultrasound evaluation of Achilles tendon will be performed. At one, two and three months after their initial evaluation, participants will receive a link to complete an online survey about their pain. Three months after their initial evaluation, a second ultrasound of Achilles tendon will be performed.

DETAILED DESCRIPTION:
At their first visit, participants will read and sign the consent form. They will then fill self-report questionnaires about their pain (using the Victorian Institute of Sport Assessment for Achilles tendinopathy score and visual analog scale) and its impact on their activities, and they will be questioned on their training habits. Then, participants will be asked to run on a treadmill for five minutes at a comfortable speed. During the run, video will be recorded to evaluate to cadence and the foot contact angle. Finally, an ultrasound of Achilles tendon will be performed to evaluate thickness, area, echogenicity and inflammation of the tendon. All the images will be revised by a physician qualified in diagnostic ultrasound and the tendinopathy will be graded according to Matthew and al. model.

One, two and three months after their initial visit, participants will receive a questionnaire by email to quantify their pain. Moreover, three months after their initial visit, participants will come back in person to the laboratory. Information about their pain, training and treatment will be collected and a second ultrasound analysis will be performed.

Statistical analysis: Baseline data will be compared using independent t-test or a Mann-Whitney U test. Significant variables in the univariate analysis will be considered as potential predictor variables. Logistic analysis regression will then be performed to identify predictive factors for pain chronicity.

ELIGIBILITY:
Inclusion Criteria:

* Have Achilles tendon pain for less than three months
* Run at least five kilometers per week
* Have a score on the Victorian Institute of Sports Assessment of Achilles tendinopathy of 80 or less
* Consent to the study

Exclusion Criteria:

* History of Achilles tendon surgery or rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Runners from Québec city region with Achilles tendon pain for less than three months
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain graded on the visual analog scale | At three months
  Pain graded on a 0 to 10 visual analog scale
Victorian Institute of Sports Assessment for Achilles tendinopathy (VISA-A) questionnaire | At three months
  Pain impact score between 0 (heavily affected) and 100 (asymptomatic)

SECONDARY OUTCOMES:
Thickness of the Achilles tendon | At three months
  Ultrasound evaluation of the tendon
Area of the Achilles tendon | At three months
  Ultrasound evaluation of the tendon
Aspect of the tendon at ultrasound evaluation graded according to Matthew and al | At three months
  Ultrasound evaluation of the tendon

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Interdisciplinary Research in Rehabilitation and Social Integration (CIRRIS), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altman AR, Davis IS. A kinematic method for footstrike pattern detection in barefoot and shod runners. Gait Posture. 2012 Feb;35(2):298-300. doi: 10.1016/j.gaitpost.2011.09.104. Epub 2011 Nov 8. PMID 22075193
- [Background] Esculier JF, Dubois B, Dionne CE, Leblond J, Roy JS. A consensus definition and rating scale for minimalist shoes. J Foot Ankle Res. 2015 Aug 19;8:42. doi: 10.1186/s13047-015-0094-5. eCollection 2015. PMID 26300981
- [Background] Matthews W, Ellis R, Furness JW, Rathbone E, Hing W. Staging achilles tendinopathy using ultrasound imaging: the development and investigation of a new ultrasound imaging criteria based on the continuum model of tendon pathology. BMJ Open Sport Exerc Med. 2020 Mar 25;6(1):e000699. doi: 10.1136/bmjsem-2019-000699. eCollection 2020. PMID 32341798